CLINICAL TRIAL: NCT07376018
Title: Adjunctive Low-carb Ketogenic Diet to Enhance Imaging-guided Neuromodulation in Treatment Resistant Depression
Brief Title: Ketogenic Diet and Neuromodulation in Treatment Resistant Depression
Acronym: ALIGN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Baszucki Group (Unknown)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6944
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD); Treatment Resistant Depression (TRD)
Keywords: Major Depressive Disorder; MDD; TRD; TMS; Glucose Control; Ketogenic Diet; Metabolic Health; Transcranial Magnetic Stimulation; iTBS; Dietary Intervention; Metabolic Psychiatry; MRS; fMRI; Intermittent Theta-Burst Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel-group interventional design in which adults with treatment-resistant depression are assigned to one of two dietary conditions (ketogenic diet or Canadian Food Guide-aligned diet) while receiving the same accelerated, connectivity-guided iTBS protocol. This design allows investigators to examine the effects of metabolic state on response to neuromodulation while holding stimulation parameters constant across groups. Both groups receive equivalent contact time with clinicians and dietitians to control for nonspecific therapeutic effects.
  The study incorporates multimodal assessments, including clinical, metabolic, and neuroimaging measures, to evaluate how changes in metabolism relate to brain network engagement and clinical response during iTBS. This structure supports both mechanistic investigation and comparison of clinical outcomes between diet conditions.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic Diet (Experimental): Participants in this arm will begin a well-formulated ketogenic diet (low carbohydrate, moderate protein, high fat) for a 3-week dietary lead-in period prior to neuromodulation, and will continue the diet for a total of 12 weeks. The diet is designed to achieve and maintain nutritional ketosis (blood ketone levels of 0.5 to 3 mmol/L). Dietitian support will be provided through scheduled counseling and ongoing monitoring using daily finger-stick ketone and glucose testing.
  Interventions: Device: Accelerated Intermittent Theta Burst Stimulation (iTBS)
- Canadian Food Guide-Aligned Diet (Active Comparator): Participants in this arm will begin a Canadian Food Guide-aligned diet for a 3-week dietary lead-in period prior to neuromodulation and will continue the diet for a total of 12 weeks. The diet will emphasize balanced intake of vegetables, fruits, whole grains, and protein foods, without specific macronutrient restrictions. Dietitian counseling will be matched in frequency and duration to the ketogenic diet arm. Nutritional monitoring will include dietary logs and metabolic assessments without targeted induction of ketosis. Participants will perform daily finger-stick glucose testing.
  Interventions: Device: Accelerated Intermittent Theta Burst Stimulation (iTBS)

INTERVENTIONS:
Device: Accelerated Intermittent Theta Burst Stimulation (iTBS) — Intermittent theta burst stimulation (iTBS), a form of repetitive transcranial magnetic stimulation (rTMS), is a non-invasive brain stimulation technique approved by the FDA and Health Canada for the treatment of TRD. In this study, participants will receive an accelerated course of image-guided, neuronavigated left dorsolateral prefrontal cortex (DLPFC) iTBS targeted based on functional connectivity with the subgenual anterior cingulate cortex (sgACC). Stimulation will consist of 600 pulses per session, delivered at 110% of resting motor threshold, with 50-minute inter-session intervals, for 8 sessions per day over 5 consecutive days.
  Other Names: repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
The goal of this clinical trial is to test whether combining a ketogenic diet (KD) with personalized, accelerated intermittent theta burst stimulation (iTBS) produces greater reductions in depressive symptoms than iTBS combined with a standard healthy diet in adults with treatment-resistant depression. The trial also aims to determine whether participants can feasibly follow a ketogenic diet during an accelerated iTBS treatment course and whether the diet produces measurable changes in ketone levels.

Specifically, the study aims to determine whether the combined intervention:

1. Reduces depressive symptoms
2. Increases circulating ketone levels
3. Is feasible and tolerable during accelerated iTBS treatment

Participants will begin either a KD or a Canadian Food Guide-aligned diet (CFGD) with a 3-week dietary lead-in period, after which they will undergo a course of personalized, accelerated iTBS while continuing their assigned diet. Before and after the iTBS treatment course, participants will complete clinical assessments, provide blood samples for metabolic testing, and undergo MRI scans to assess brain connectivity. Ketone levels will be measured daily throughout the 12-week dietary intervention. Within-group and between-group differences will be compared to characterize changes in clinical outcomes, metabolism, and brain functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 of any sex, gender identity, ethnicity and socioeconomic status
* Currently experiencing a major depressive episode as defined by DSM-5-TR criteria and confirmed by a study physician
* Presenting with at least moderate symptom severity (MADRS ≥ 20)
* Meeting criteria for treatment-resistant depression (TRD), defined as non-response to at least two adequate antidepressant trials
* Neuromodulation-naïve (no past rTMS or electroconvulsive therapy)
* Able to provide informed consent
* Available for the 15-week intervention and willing to follow either a ketogenic or Canadian Food Guide-aligned diet

Exclusion Criteria:

* Medical/psychiatric co-morbidities that prevent participation in the study or where depression is not the primary psychiatric symptom of concern
* History of epilepsy, stroke, or major neurological conditions, psychosis, or substance dependence within the last 6 months
* Physical or cognitive disability interfering with participation
* Females who are pregnant (self-report or via blood work), nursing, or planning a pregnancy during the timespan of the study BMI < 20 kg/m²
* Suicide attempts in the past 12 months
* Active suicidal intent as confirmed by study psychiatrist
* Active eating disorder in the past 12 months
* Currently following a KD
* Habitual low-carb diet in the past 6 months
* GI disorders or food allergies incompatible with dietary protocols
* Alcohol use >3 drinks/day or >14/week
* Use of anticonvulsants (benzodiazepines with a dose of <2 lorazepam equivalents will be permitted), GABA agonists, or medications reducing TMS efficacy
* Serious medical illness
* Contraindications to MRI
* Unwillingness to perform daily finger-stick testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Score on the Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Change in depression symptomatology as assessed by the clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) (range 0-60). Higher scores indicate worse outcomes (greater severity of depressive symptoms)
Changes in Ketone Levels | Baseline through week 12
  Change in fasting morning β-hydroxybutyrate concentrations over the treatment period relative to baseline. Fasting β-hydroxybutyrate will be measured daily via finger-stick ketone testing, and longitudinal change will be analyzed across the treatment period.
Safety and Tolerability | Baseline through week 12
  Frequency, severity, and relatedness of adverse events and clinically significant laboratory abnormalities, and discontinuations due to adverse effects, with specific attention to KD-related effects (e.g., hypoglycemia, dehydration, electrolyte disturbances, gastrointestinal symptoms, dyslipidemia) and mood destabilization/suicidality.

SECONDARY OUTCOMES:
Changes in ¹H-MRS Neurochemical Metabolites | Baseline to Week 4 (post-iTBS)
  Proton magnetic resonance spectroscopy will quantify changes in metabolites associated with neuroplasticity and metabolic function. Metabolite concentrations will be compared from baseline to post-treatment to determine whether nutritional ketosis enhances neurochemical responses to iTBS.
Changes in Resting-State Functional Connectivity | Baseline to Week 4 (post-iTBS)
  Resting-state fMRI will be used to assess changes in intrinsic functional connectivity within fronto-cingulate and fronto-striatal networks. Connectivity between the individualized DLPFC stimulation target and the subgenual anterior cingulate cortex will be quantified. Baseline-to-post-treatment changes will be used to evaluate diet-related enhancement of iTBS-induced network modulation.
Changes in Task-Evoked Brain Activation | Baseline to Week 4 (post-iTBS)
  Task-based fMRI will be used to measure changes in activation within predefined mood-regulation circuits. Contrast maps from an emotional processing task will be compared from baseline to post-treatment to assess neural circuit engagement associated with iTBS combined with dietary intervention.
Changes in Metabolic Biomarkers | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Changes in fasting metabolic and inflammatory biomarkers across the study period. Biomarkers include HbA1C, fasting glucose, lipid profile, total protein, albumin, total bilirubin, ALT, AST, ALP, electrolytes, urea, calcium, BDNF, IL-6, TNF-α, and C-reactive protein (CRP), with pregnancy testing (hCG) in females where applicable.
Change in Secondary Depression Scores | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Baseline grid-version of the 17-item Hamilton Depression Rating Scale (HDRS) score. The HDRS is a 17-item clinician-administered rating scale designed to assess severity of depressive symptoms. The score range is 0 to 52, with higher score indicating more severe depression.
Change in Self-Reported Depressive Symptoms | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Self-reported depressive symptom severity will be assessed using the PHQ-9 with changes measured from baseline to each assessment point through the end of treatment. Higher scores on the PHQ-9 (0-27) represent greater depressive severity.
Functional Disability | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Functional disability will be measured using the WHODAS 2.0, with changes evaluated from baseline to the end of treatment. Higher WHODAS scores indicate greater impairment.
Well-being | Baseline, Day (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Well-being will be evaluated using the WHO-5 Well-Being Index, measured from baseline to the end of treatment. Higher WHO-5 scores represent better well-being.
Change in Anxiety Measure | Baseline, Day (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Anxiety symptom severity will be assessed using the Generalized Anxiety Disorder-7 (GAD-7), with improvement examined from baseline to the end of treatment. Higher GAD-7 scores reflect more severe anxiety
Anthropometric Outcomes | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Anthropometric outcomes, including BMI, waist circumference, and waist-to-hip ratio, will be recorded to evaluate changes in adiposity and fat distribution from baseline to the end of treatment. Higher waist-to-hip ratios indicate greater central adiposity.
Physiological Measures | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Resting systolic/diastolic blood pressure and heart rate will be measured to assess physiological changes. Higher blood pressure values reflect worse cardiovascular status.
Executive Functioning | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Executive functioning will be assessed using the NIH Toolbox Dimensional Change Card Sort Test and the Flanker Inhibitory Control and Attention Test, with changes evaluated from baseline to the end of treatment. Higher scores reflect better cognitive performance.
Working Memory | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Working memory will be measured using the NIH Toolbox List Sorting Working Memory Test, with changes compared from baseline to post-treatment. Higher scores indicate stronger working memory ability.
Episodic Memory | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Episodic memory will be assessed using the NIH Toolbox Auditory Verbal Learning Test and the Picture Sequence Memory Test, with changes evaluated from baseline to the end of treatment. Higher scores indicate better episodic memory performance.
Processing Speed | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Processing speed will be evaluated using the NIH Toolbox Oral Symbol Digit Test and the Pattern Comparison Processing Speed Test, with changes assessed from baseline to post-treatment. Higher scores reflect faster processing speed.
Treatment Expectancy | Baseline
  Treatment expectancy will be assessed using the Stanford Expectations of Treatment Scale (SETS), administered at baseline to evaluate participants' expectations prior to the intervention. Higher scores on the SETS indicate stronger positive treatment expectancy.
Perceived Physical Capacity | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  The modified Rating of Perceived Exertion (RPE) scale will be used to assess participants' perceived physical effort and tolerance during routine physical activities and daily tasks. This subjective measure captures how hard the body feels it is working based on internal sensations such as breathing, cardiovascular strain, muscle fatigue, and overall exertion, providing an index of perceived functional capacity for physical activity.
Objective Physical Capacity | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Objective indices of physical capacity and fatigue will be obtained using handgrip dynamometry. Maximal voluntary force (MVF) will be measured as the average of three maximal-effort trials, reflecting peak isometric grip strength and overall neuromuscular capacity of the hand and forearm muscles.
Fatigue | Baseline, Day 5 (post-iTBS), Week 4 (post-iTBS), Week 8 (post-iTBS)
  Time to exhaustion (TTE) during a sustained submaximal grip task will be used to quantify fatigue resistance and endurance, defined as the duration for which participants can maintain a prescribed grip force before they are unable to sustain the target level.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and relevant supporting documentation (including the study protocol, statistical analysis plan, and data dictionary) will be shared to enable secondary research. Data will be shared with qualified researchers for scientifically sound analyses, subject to approval and execution of a data use agreement in accordance with Sunnybrook Research Institute policies. Requests for access will be reviewed to ensure scientific merit, feasibility, and protection of participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol and informed consent form will be published prior to study initiation. Trial results will be disseminated as soon as feasible after study completion. De-identified IPD will be available beginning 12 months after publication of the primary results (or 12 months after study completion if no publication occurs).
Access Criteria: Shared data will include de-identified IPD and supporting documents (study protocol, statistical analysis plan, and data dictionary).
  Access will be limited to researchers with appropriate institutional affiliation and documented ethics approval, who submit a methodologically sound proposal. Requests will be reviewed by the study Principal Investigator (or designated data access committee).
  Approved users will obtain access through secure, institutionally approved data-sharing systems. All users must sign a data use agreement that prohibits re-identification, onward sharing, and any use outside the approved proposal.